CLINICAL TRIAL: NCT00909415
Title: Urodynamic Evaluation in Patients With Anorectal Malformation According to Spinal Cord Abnormalities
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2009-0171
Record Dates: First submitted 2009-05-26; First posted 2009-05-28 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Anorectal Malformation
Keywords: patients with anorectal malformation
MeSH Terms: conditions — Anorectal Malformations

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This study will examine the effects of spinal cord abnormalities on perioperative neurovesical dysfunction in patients with anorectal abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Anorectal malformation patients who underwent preoperative and postoperative urodynamic studies

Exclusion Criteria:

* Severe artifacts in urodynamic result graph when the postoperative urodynamic study was done after spinal surgery

Ages: 1 Month to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with anorectal malformation
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea